CLINICAL TRIAL: NCT03764293
Title: A Randomized, Open-Label, International, Multi-Center, Phase 3 Clinical Study of PD-1 Antibody SHR-1210 Plus Apatinib Mesylate Versus Sorafenib as First-Line Therapy in Patients With Advanced Hepatocellular Carcinoma (HCC) Who Have Not Previously Received Systemic Therapy
Brief Title: A Study to Evaluate SHR-1210 in Combination With Apatinib as First-Line Therapy in Patients With Advanced HCC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-III-310
Record Dates: First submitted 2018-11-28; First posted 2018-12-05 (Actual); Results first posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2023-02

CONDITIONS: Locally Advanced or Metastatic and Unresectable HCC
MeSH Terms: conditions — Neoplasm Metastasis | interventions — camrelizumab; apatinib; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SHR-1210 (Experimental): SHR-1210+Apatinib
  Interventions: Drug: SHR-1210; Drug: Apatinib
- Control (Active Comparator): Sorafenib
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: SHR-1210 — Subjects receive SHR-1210 intravenously, Dosage form: lyophilised powder, Strength: 200 mg /vial
  Other Names: Camrelizumab
  Arms: SHR-1210
Drug: Apatinib — Subjects receive Apatinib orally, Dosage form: tablet, Strength: 250 mg/tablet
  Other Names: Rivoceranib
  Arms: SHR-1210
Drug: Sorafenib — Subjects receive Sorafenib orally, Dosage form: tablet, Strength: 0.2 g/tablet
  Arms: Control

SUMMARY:
This is a randomized, open-label, international, multi-center, phase III trial to evaluate the efficacy and safety of SHR-1210 plus apatinib mesylate versus sorafenib as first-line therapy in patients with advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically or cytologically confirmed advanced HCC
* No previous systematic treatment for HCC
* Have at least one measurable lesion (in accordance with RECIST v1.1)
* BCLC stage B or C, and not suitable for surgical or local therapy, or has progressed following surgical and/or local therapy
* ECOG-PS score 0 or 1
* Child-Pugh Class: Grade A
* Life Expectancy of at least 12 weeks
* Subjects with HBV infection: HBV DNA<500 IU/ml or < 2500 copy/mL, and have received anti-HBV therapy for at least 14 days prior to enrollment in the study
* Subjects with HCV-RNA(+) must receive antiviral therapy
* Adequate organ function

Exclusion Criteria:

* Known hepatocholangiocarcinoma, sarcomatoid HCC, mixed cell carcinoma and lamellar cell carcinoma; other active malignant tumor except HCC within 5 years or simultaneously
* Moderate-to-severe ascites with clinical symptoms
* History of gastrointestinal hemorrhage within 6 months prior to the start of study treatment or clear tendency of gastrointestinal hemorrhage
* Abdominal fistula, gastrointestinal perforation or intraperitoneal abscess within 6 months prior to the start of study treatment
* Known genetic or acquired hemorrhage or thrombotic tendency
* Thrombosis or thromboembolic event within 6 months prior to the start of study treatment
* Cardiac clinical symptom or disease that is not well controlled
* Hypertension that can not be well controlled through antihypertensive drugs
* Factors to affect oral administration
* History of hepatic encephalopathy
* Previous or current presence of metastasis to central nervous system
* HIV infection
* Combined hepatitis B and hepatitis C co-infection
* Be ready for or previously received organ or allogenic bone marrow transplantation
* Interstitial lung disease that is symptomatic or may interfere with the detection and management of suspected drug-related pulmonary toxicity
* Active known, or suspected autoimmune disease
* Subjects with a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days of first administration of study treatment
* Use of potent CYP3A4 inducers or inhibitors within 2 weeks prior to the signature of ICF
* Known history of serious allergy to any monoclonal antibody or targeted anti-angiogenic drug
* Severe infection within 4 weeks prior to the start of study treatment
* Palliative radiotherapy for non-target lesions to control symptoms is allowed, but it must be completed at least 2 weeks prior to the start of study treatment
* Treatment of other investigational product(s) within 28 days prior to the start of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2023-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shukui Qin, MD, Principal Investigator — Eastern Theater General Hospital,QinHuai District Medical Area
Locations (121):
- United States (8):
  - Beverly Hills Cancer Center, Beverly Hills, California
  - University of California San Diego (UCSD)-Moores Cancer Center, La Jolla, California
  - University of California - Irvine, Orange, California
  - University of Maryland, Baltimore, Maryland
  - Cornell University Weill Cornell Medical College, New York, New York
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Renovatio Clinical, The Woodlands, Texas
- Belgium (5):
  - Cliniques Universitaires de Bruxelles Hopital Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZA, Edegem
  - AZ Maria Middelares, Ghent
  - AZ Groeninge, Kortrijk
- China (37):
  - Anhui Provincal Cancer Hospital, Hefei, Anhui
  - Anhui Provincal Hospital, Hefei, Anhui
  - The First Affiliated Hospital Of Anhui Medical University, Hefei, Anhui
  - The Second Affiliated Hospital Of Anhui Medical University, Hefei, Anhui
  - Chinese Academy of Medical Sciences Cancer Hospital, Beijing, Beijing Municipality
  - Beijing cancer Hospital, Beijing, Beijing Municipality
  - Peking University International Hospital, Beijing, Beijing Municipality
  - The Second Hospital Affiliated To AMU, Chongqing, Chongqing Municipality
  - The First Hospital Affiliated To AMU, Chongqing, Chongqing Municipality
  - TheThird Affiliated Hospital ,Army Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of ChongQing Medical University, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The 940th Hospital of the joint logistic support force of People's Liberation Army, Lanzhou, Gansu
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - NanFang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The first affiliated hospital of guangxi medical university, Nanning, Guangxi
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Wuhan Union Hospital,Tongji Medical College,Huazhong University of Science&Technology, Wuhan, Hubei
  - Tongji hospital,Tongji Medical College,Huazhong University of Science&Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Eastern Theater General Hospital, Qinhuai District Medical Area, Nanjing, Jiangsu
  - The First Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Sixth People's Hospital of Shengyang, Shengyang, Liaoning
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Shandong Cancer Hospital Affiliated to Shandong University, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Sichuan Cancer Hospital&Institute, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - ZheJiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
- Charite Universitaetsmedizin Berlin - Campus Virchow-Klinikum Berlin, Berlin, Germany
- Hong Kong (4):
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - The University of Hong Kong, Hong Kong
  - Tuen Mun Hospital, Hong Kong
  - The Chinese University of Hong Kong, Shatin
- Italy (8):
  - A.S.L. Napoli 1 Centro Ospedale del Mare, Ponticelli, Napoli
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi IRCCS, Bologna
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Presidio Spedali Civili), Brescia
  - Azienda Ospedaliero-Universitaria, Cagliari
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Azienda Ospedaliera Universitaria Integrata Verona (Ospedale Borgo Roma), Verona
- Poland (8):
  - Centrum Medyczne Pratia Gdynia, Gdynia
  - Centrum Onkologii-Instytut im.M.Sklodowskiej Curie, Gliwice
  - Pratia MCM Krakow, Krakow
  - Przychodnia Med-Polonia Sp. z o.o., Poznan
  - Wielkopolskie Centrum Onkologii, Poznan
  - Centrum Zdrowia MDM, Warsaw
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie - Państwowy Instytut Badawczy, Warsaw
  - NZOZ Centrum Badan Klinicznych, Wroclaw
- Russia (13):
  - SBIH of Arkhangelsk region "Arkhangelsk Clinical Oncological Dispensary", Arkhangelsk
  - SBHI Chelyabinsk Regional Clinical Center for Oncology and Nuclear Medicine, Chelyabinsk
  - Irkutsk Regional Oncology Dispensary, Irkutsk
  - SBIH " Clinical Oncological Dispensary # 1", Krasnodar
  - RBIH "Kursk regional clinical oncology dispensary" of Kursk Region Healthcare Committee, Kursk
  - "VitaMed" LLC, Moscow
  - SBIH of Moscow city "Moscow city oncology hospital №62" of Moscow Healthcare departement, Moscow
  - CJSC Avicenna, Novosibirsk
  - BHI of Omsk region "Clinical Oncology Dispensary", Omsk
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - SPb SBIH "City Clinical Oncological Dispensary", Saint Petersburg
  - FBI "Scientific Research Institute of Oncology n. a. N. N. Petrov", Saint Petersburg
  - SBIH Republican Clinical Oncological Dispensary of the MoH of Republic Bashkortostan, Ufa
- South Korea (8):
  - Seoul National University Bundang Hospital Gyeonggi-do, Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Dong-A University Hospital, Busan
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (7):
  - Hospital Universitario Reina Sofia, Córdoba, Córdoba
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario HM Madrid Sanchinarro, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- Taiwan (8):
  - Changhua Christian Medical Foundation Changhua Christian Hospital, Changhua
  - Chang Gung Memorial Hospital, Chiayi, Chiayi City
  - E-DA Cancer Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District
- Turkey (Türkiye) (6):
  - Baskent University Adana Application and Research Center, Adana
  - Dr. Abdurrahman Yurtaslan Oncology Teaching and Research Hospital, Ankara
  - Ankara City Hospital, Ankara
  - Istanbul University Cerrahpasa - Cerrahpasa Medical Faculty, Istanbul
  - Bakirkoy Dr. Sadi Konuk Teaching and Research Hospital, Istanbul
  - Inonu Uni. Med. Fac., Malatya
- Ukraine (8):
  - CNE"City Clin Hosp#4"of Dnipro City Council Dept of Chemotherapy SI Dnipropetrovsk MA of MOHU, Dnipro
  - Communal Non-profit Enterprise Regional Center of Oncology, Kharkiv
  - CI of Healthcare Regional Clinical Specialized Dispensary of the Radiation Protection, Kharkiv
  - Medical Center of Limited Liability Company Medical Center Concilium Medical, Kyiv
  - Communal Enterprise Volyn Regional Medical Center of Oncology of Volyn Regional Council, Lutsk
  - Communal Institution Odesa Regional Clinical Hospital, Odesa
  - CNCE of SRC Sumy Reg Clinical Oncology Dispensary, SSU, Chair of Oncology and Radiology, Sumy
  - Zaporizhzhya City Clinical Hospital #3, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qin S, Gu S, Chan SL, Bai Y, Ren Z, Lin X, Chen Z, Jia W, Jin Y, Guo Y, Hu X, Meng Z, Liang J, Xiong J, Ren H, Yang F, Li W, Chen Y, Zeng Y, Xu L, Yuan X, Li D, Sultanbaev A, Pazgan-Simon M, Pisetska M, Melisi D, Ponomarenko D, Du J, Shi W, Cheng AL, Kaseb A, Vogel A; CARES-310 Study Group. Camrelizumab plus rivoceranib versus sorafenib as first-line therapy for unresectable hepatocellular carcinoma (CARES-310): final analysis of a randomised, open-label, international, phase 3 study. Lancet Oncol. 2025 Dec;26(12):1598-1611. doi: 10.1016/S1470-2045(25)00543-1. PMID 41308676
- [Derived] Qin S, Chan SL, Gu S, Bai Y, Ren Z, Lin X, Chen Z, Jia W, Jin Y, Guo Y, Hu X, Meng Z, Liang J, Cheng Y, Xiong J, Ren H, Yang F, Li W, Chen Y, Zeng Y, Sultanbaev A, Pazgan-Simon M, Pisetska M, Melisi D, Ponomarenko D, Osypchuk Y, Sinielnikov I, Yang TS, Liang X, Chen C, Wang L, Cheng AL, Kaseb A, Vogel A; CARES-310 Study Group. Camrelizumab plus rivoceranib versus sorafenib as first-line therapy for unresectable hepatocellular carcinoma (CARES-310): a randomised, open-label, international phase 3 study. Lancet. 2023 Sep 30;402(10408):1133-1146. doi: 10.1016/S0140-6736(23)00961-3. Epub 2023 Jul 24. PMID 37499670

RESULTS

PARTICIPANT FLOW:
Groups:
- Camrelizumab+Rivoceranib Arm: Camrelizumab+rivoceranib arm: Rivoceranib 250 mg orally, QD, within 30 minutes after a meal, continuously.
  Camrelizumab 200 mg IV infusion, over 30 minutes, Q2W. The interval between two doses should not be less than 12 days.
- Sorafenib Arm: Sorafenib arm: Sorafenib 400 mg orally, BID, in a fasted state (at least 1 hour before or 2 hours after a meal), continuously.
Period: Overall Study
Arm/Group | Camrelizumab+Rivoceranib Arm | Sorafenib Arm
Started | 272 | 271
Treated | 272 | 269
Completed | 230 | 249
Not Completed | 42 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Camrelizumab+Rivoceranib Arm | Sorafenib Arm | Total
Number analyzed (Participants) | 272 | 271 | 543
Age, Customized [Number; unit: participants]
  <65 Years | 191 | 210 | 401
  >=65 Years | 81 | 61 | 142
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 41 | 86
  Male | 227 | 230 | 457
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 226 | 224 | 450
  Black Or African American | 1 | 0 | 1
  White | 44 | 46 | 90
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death from any cause.
Time Frame: Up to approximately 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Camrelizumab+Rivoceranib Arm | Sorafenib Arm
Number analyzed (Participants) | 272 | 271
months | 22.1 [19.1 to 27.2] | 15.2 [13.0 to 18.5]

2. Primary Outcome: Progression-free Survival (PFS) Evaluated by the Blinded Independent Review Committee (BIRC) Based on RECIST v1.1
Description: PFS was defined as the time from randomization to the first occurrence of progressive disease (PD) by tumor image evaluation or death from any cause whichever occurs first as determined by BIRC according to RECIST v1.1. PD: at least a 20% increase in the sum of diameters of target lesions and the sum of diameters must also demonstrate an absolute increase of >/= 5 millimeters (mm), or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to approximately 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Camrelizumab+Rivoceranib Arm | Sorafenib Arm
Number analyzed (Participants) | 272 | 271
months | 5.6 [5.5 to 7.4] | 3.7 [3.1 to 3.7]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR defined as the percentage of subjects with complete response (CR) or partial response (PR) evaluated by the BIRC or investigator based on RECIST v1.1. CR: disappearance of all target lesions. PR: At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. Overall Response (OR)=CR+PR.
Time Frame: Up to approximately 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Camrelizumab+Rivoceranib Arm | Sorafenib Arm
Number analyzed (Participants) | 272 | 271
percentage of participants | 25 [20 to 31] | 6 [3 to 9]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR defined as the percentage of subjects with complete response, partial response or stable disease (SD) ≥ 8 weeks evaluated by the BIRC or investigator based on RECIST v1.1. Complete response (CR) was defined as Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response (PR) was defined as at least a 30% decrease in the sum of the diameter of TL, taking as reference the baseline sum of diameters. Stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Up to approximately 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Camrelizumab+Rivoceranib Arm | Sorafenib Arm
Number analyzed (Participants) | 272 | 271
percentage of participants | 78 [73 to 83] | 54 [48 to 60]

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR defined as time from the date of first record of objective response (CR or PR) to the first occurrence of radiological progression or death, whichever comes first, evaluated by the BIRC or investigator based on RECIST v1.1. Complete response (CR) was defined as Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response (PR) was defined as at least a 30% decrease in the sum of the diameter of TL, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Camrelizumab+Rivoceranib Arm | Sorafenib Arm
Number analyzed (Participants) | 272 | 271
months | 14.8 [8.4 to NA] — NA=the 75-percentile DOR is not reached and hence the upper limit of the 95% CI of the median DOR is not estimable due to a lot of censoring and not enough disease progressions/events. | 9.2 [5.3 to NA] — NA=the 75-percentile DOR is not reached and hence the upper limit of the 95% CI of the median DOR is not estimable due to a lot of censoring and not enough disease progressions/events.

ADVERSE EVENTS:
Time Frame: Up to approximately 3 years
Arm/Group | Camrelizumab+Rivoceranib Arm | Sorafenib Arm
All-Cause Mortality (participants affected / at risk) | 34/272 | 17/269
Serious Adverse Events (participants affected / at risk) | 114/272 | 49/269
Other Adverse Events (participants affected / at risk) | 268/272 | 262/269
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Camrelizumab+Rivoceranib Arm (N=272) | Sorafenib Arm (N=269)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 12 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 4
Ascites (Gastrointestinal disorders) | 4 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Immune-mediated enterocolitis (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Gastriculcer (Gastrointestinal disorders) | 1 | 0
Immune-mediated pancreatitis (Gastrointestinal disorders) | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 4
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Anal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Urethral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 10 | 2
Alanine aminotransferase increased (Investigations) | 8 | 1
Blood bilirubin increased (Investigations) | 8 | 2
Platelet count decreased (Investigations) | 5 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0
Bilirubin conjugated increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 4 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 3 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Biliary obstruction (Hepatobiliary disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 2
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0
Biloma (Hepatobiliary disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 10 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Immune-mediated encephalitis (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Myasthenic syndrome (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 2
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 0
COVID-19 (Infections and infestations) | 2 | 1
Sepsis (Infections and infestations) | 2 | 2
Abdominal sepsis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Periodontitis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 2
Peritonitis bacterial (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 2
Biliary tract infection (Infections and infestations) | 0 | 1
Colonic abscess (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Pyrexia (General disorders) | 4 | 2
Death (General disorders) | 2 | 0
Multiple organ dysfunction syndrome (General disorders) | 2 | 1
Asthenia (General disorders) | 1 | 1
Pain (General disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2
Cardiac failure (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Immune-mediated myocarditis (Cardiac disorders) | 1 | 0
Reactive capillary endothelial proliferation (Immune system disorders) | 4 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Affective disorder (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Camrelizumab+Rivoceranib Arm (N=272) | Sorafenib Arm (N=269)
Anaemia (Blood and lymphatic system disorders) | 71 | 48
Hypothyroidism (Endocrine disorders) | 59 | 20
Diarrhoea (Gastrointestinal disorders) | 90 | 114
Nausea (Gastrointestinal disorders) | 45 | 22
Abdominal distension (Gastrointestinal disorders) | 36 | 18
Abdominal pain upper (Gastrointestinal disorders) | 32 | 15
Vomiting (Gastrointestinal disorders) | 30 | 18
Abdominal pain (Gastrointestinal disorders) | 29 | 33
Constipation (Gastrointestinal disorders) | 24 | 20
Gingival bleeding (Gastrointestinal disorders) | 21 | 16
Ascites (Gastrointestinal disorders) | 17 | 16
Stomatitis (Gastrointestinal disorders) | 17 | 10
Toothache (Gastrointestinal disorders) | 14 | 8
Fatigue (General disorders) | 68 | 34
Pyrexia (General disorders) | 45 | 32
Asthenia (General disorders) | 37 | 23
Oedema peripheral (General disorders) | 25 | 4
Reactive capillary endothelial proliferation (Immune system disorders) | 79 | 1
Upper respiratory tract infection (Infections and infestations) | 26 | 15
Aspartate aminotransferase increased (Investigations) | 178 | 137
Alanine aminotransferase increased (Investigations) | 154 | 115
Platelet count decreased (Investigations) | 138 | 105
Blood bilirubin increased (Investigations) | 131 | 112
Gamma-glutamyltransferase increased (Investigations) | 88 | 80
White blood cell count decreased (Investigations) | 79 | 48
Neutrophil count decreased (Investigations) | 78 | 33
Weight decreased (Investigations) | 67 | 70
Blood alkaline phosphatase increased (Investigations) | 63 | 56
Bilirubin conjugated increased (Investigations) | 53 | 52
Blood bilirubin unconjugated increased (Investigations) | 40 | 33
Blood lactate dehydrogenase increased (Investigations) | 38 | 37
Lymphocyte count decreased (Investigations) | 29 | 23
Amylase increased (Investigations) | 28 | 13
Blood thyroid stimulating hormone increased (Investigations) | 26 | 8
Total bile acids increased (Investigations) | 25 | 11
Urinary occult blood positive (Investigations) | 25 | 12
Lipase increased (Investigations) | 22 | 13
Occult blood positive (Investigations) | 22 | 20
Electrocardiogram QT prolonged (Investigations) | 19 | 10
Blood creatinine increased (Investigations) | 16 | 7
Hypoalbuminaemia (Metabolism and nutrition disorders) | 84 | 62
Decreased appetite (Metabolism and nutrition disorders) | 58 | 46
Hypokalaemia (Metabolism and nutrition disorders) | 45 | 34
Hyponatraemia (Metabolism and nutrition disorders) | 34 | 22
Hyperglycaemia (Metabolism and nutrition disorders) | 32 | 15
Hypophosphataemia (Metabolism and nutrition disorders) | 26 | 48
Hypocalcaemia (Metabolism and nutrition disorders) | 20 | 8
Hyperuricaemia (Metabolism and nutrition disorders) | 11 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 36 | 22
Headache (Nervous system disorders) | 39 | 7
Dizziness (Nervous system disorders) | 20 | 6
Insomnia (Psychiatric disorders) | 14 | 12
Proteinuria (Renal and urinary disorders) | 136 | 82
Haematuria (Renal and urinary disorders) | 38 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 31 | 14
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 26 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 | 8
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 101 | 163
Rash (Skin and subcutaneous tissue disorders) | 51 | 55
Pruritus (Skin and subcutaneous tissue disorders) | 21 | 13
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 52
Hypertension (Vascular disorders) | 190 | 118

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All clinical study findings and documents will be regarded as confidential. The investigator and members of his/her research team must not disclose such information without prior written approval from the sponsor.

DOCUMENTS (2):
  • Study Protocol (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/93/NCT03764293/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/93/NCT03764293/SAP_001.pdf